CLINICAL TRIAL: NCT02953288
Title: Differential Diagnosis and Clinical Treatment Strategies of Thyroid Nodules.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Department of Endocrinology, Shanghai 10th People's Hospital
Other Study IDs: Research center of the thyroid
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Thyroid tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Benign thyroid nodules: Benign thyroid nodules
- Thyroid Carcinoma: Thyroid Carcinoma

SUMMARY:
To investigate the genetic mutations of patients with thyroid carcinoma and find molecular targets for therapy.

DETAILED DESCRIPTION:
In previous studies, we have found highly prevalent TERT promoter mutations in aggressive thyroid cancers. So we plan to perform further research to investigate the genetic mutations of patients with thyroid carcinoma and find molecular targets for therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with thyroid nodule

Exclusion Criteria:

* Coagulant function abnormality
* pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with thyroid nodule
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Gene sequencing | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Study Director — Sanghai Tenth People's Hospital, Shanghai, China
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided